CLINICAL TRIAL: NCT03345394
Title: Effectiveness of Contingency Management in the Treatment of Crack Addiction for Individuals Living in the "Crackland" Region. A Single-blind Randomized Controlled Trial
Brief Title: Effectiveness of Contingency Management in the Treatment of Crack Addiction in Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Washington State University (Other)
Responsible Party: Principal Investigator, André de Queiroz Constantino Miguel, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAPESP 2017/05371-8
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Substance Use Disorders; Contingency Management; Addiction, Cocaine
Keywords: crack cocaine; contingency management; ambulatory treatment; Brazil
MeSH Terms: conditions — Substance-Related Disorders; Cocaine-Related Disorders

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial
Who Masked: Investigator
Masking Description: researchers had no contact with participants during the 12 week trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (Active Comparator): 12 weeks of standard treatment offered by Unidade Recomeço Helvétia treatment program
  Interventions: Behavioral: Standard treatment
- Contingency Management (Experimental): 12 weeks of standard treatment offered at Unidade Recomeço Helvétia treatment program associated with Contingency Management
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Participants will receive vouchers with monetary value for submitting crack cocaine negative urine samples
  Arms: Contingency Management
Behavioral: Standard treatment — Participants will receive the standard treatment offered at Unidade Recomeço Helvétia treatment program
  Arms: Standard Treatment

SUMMARY:
Crack addiction has become a severe public health problem in Brazil. Crack users present elevated prevalence rates of psychiatric comorbidities, sexual transmitted infections and unemployment with high probability of living or have lived in the streets, history of incarceration and engagement in illegal activities. For the last 20 years a treatment called Contingency Management (CM) have achieved the best results regarding reduction of substance use, promotion of abstinence, treatment attendance and retention in treatment. The first CM study conducted in Brazil advocates for the efficacy of CM on all of these outcomes, suggesting that CM can be effective in a Brazilian population of crack users.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effectiveness of Contingency Management (CM) for crack users living in the "Crackland" region. To achieve this goal, regular treatment staff from Unidade Recomeço Helvétia treatment service will be capacitated in CM to latter-on apply the CM intervention in their respective services. The design will be a single-blind randomized clinical trial composed of a sample of 100 subjects with current diagnose for crack/cocaine dependence. Participants allocated to the control condition will receive 12 weeks of the usual care treatment provided by these two treatment facilities. Participants allocated to the experimental condition will receive the exact same treatment as control participants associated with CM. CM procedure will occur 2 timer per week (every Monday and Thursday or Tuesday and Friday). Primary outcomes are: (1)retention in treatment; (2) reduction of crack use; (3) promotion of continuous crack cocaine abstinence. Secondary findings are reduction on psychiatric symptomatology. The investigator hypothesis is that participants in the CM condition will have a better treatment response in all studied outcomes.

ELIGIBILITY:
Inclusion Criteria:

* DSM-V diagnose for crack cocaine use disorder

Exclusion Criteria:

* being under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre M de Queiroz Constantino Miguel, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Unidade Recomeço Helvétia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Treatment | Contingency Management
Started | 48 | 50
Completed | 48 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: all participants enrolled in the study were analyzed (intention to treat)
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Contingency Management | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (9.2) | 37.2 (9) | 38.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 40 | 43 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 27 | 53
  White | 21 | 22 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 48 | 50 | 98
Negative urine exam at baseline [Count of Participants; unit: Participants] | 28 | 22 | 50

OUTCOME MEASURES:

1. Primary Outcome: Pattern of Crack Cocaine Use
Description: Percentage of negative crack cocaine urine samples submitted during the 12 weeks of treatment
Time Frame: 12 weeks
Population: all enrolled participants were analyzed (intention to treat)
Measure: Mean (Standard Deviation); unit: percent of negative cocaine samples
Arm/Group | Standard Treatment | Contingency Management
Number analyzed (Participants) | 48 | 50
percent of negative cocaine samples | 14.3 (4.6) | 40.7 (5.8)

2. Primary Outcome: Promotion of Continuous Crack Cocaine Abstinence
Description: Longest duration of continuous abstinence achieved (in weeks)
Time Frame: 12 weeks
Population: all participants enrolled in the study were analyzed (intention to treat)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Standard Treatment | Contingency Management
Number analyzed (Participants) | 48 | 50
weeks | 1.5 (3.4) | 4.35 (4.7)

3. Secondary Outcome: Treatment Retention
Description: time elapsed between treatment entry and last time present in treatment (in weeks)
Time Frame: 12 weeks
Population: all participants enrolled in the study where analyzed (intention to treat)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Standard Treatment | Contingency Management
Number analyzed (Participants) | 48 | 50
weeks | 3.4 (4.8) | 7 (5.2)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Because this study did not include a pharmacological intervention, the only adverse event information collected was mortality.
Arm/Group | Standard Treatment | Contingency Management
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT03345394/Prot_SAP_000.pdf